CLINICAL TRIAL: NCT02610049
Title: Randomized, Controlled Trial of Art Therapy During Cognitive Processing Therapy for PTSD
Brief Title: Trial of Art Therapy During Cognitive Processing Therapy for PTSD
Acronym: Art_Tx_PTSD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator has retired.
Sponsor: Hampton VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-04
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Post-traumatic Stress Disorder; Stress Disorder, Post-Traumatic
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole; Reproductive Techniques, Assisted; Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Subjects will receive 8 sessions of Cognitive Processing Therapy.
  Interventions: Behavioral: Cognitive Processing therapy
- Experimental (Experimental): Subjects will receive 8 sessions of CPT + Art Therapy 8 sessions of individual therapy.
  Interventions: Behavioral: Art + CPT
- Experimental 2 (Experimental): Subject to receive 8 sessions of individual therapy for Art + CPT Cognitive Processing Therapy intervention pre-specified to be administered separately.
  Interventions: Behavioral: CPT + Art Therapy

INTERVENTIONS:
Behavioral: Cognitive Processing therapy — 8 sessions of standard CPT from CPT manual developed by Dr. S Resick, Monson & Chard (11/2010)
  Other Names: CPT
  Arms: Control
Behavioral: Art + CPT — 8 sessions of individual therapy of mixes techniques Art + CPT 8 sessions of standard CPT (same 8 as in control group) from manual developed by Dr.s Resick, Monson & Chard (11/2010)
  Arms: Experimental
Behavioral: CPT + Art Therapy — Subjects to complete 8 sessions of standard Cognitive Processing Therapy from manual developed by Dr. S. Resick, Monson & Chard (1/2010) CPT + Art Therapy of mixed individual techniques
  Arms: Experimental 2

SUMMARY:
This is a randomized, controlled trial of adjunctive art therapy during cognitive processing therapy for PTSD.

DETAILED DESCRIPTION:
The objective of this study is to examine the effects of art therapy with combat veterans who have PTSD and to measure if it reduces symptoms more than verbal Cognitive Processing Therapy (CPT) alone. This study will incorporate art processes and materials into an already established protocol of CPT in order to create a sense of safety for veterans in beginning therapy, and access the nonverbal parts of the trauma in order to process it. Art-making will be used to help veterans address trauma and integrate who they were before the trauma with who they are currently. It will assist in addressing the grief and loss caused by combat, and will be used as veterans begin building a worldview and self-concept that are not filled with trauma and war. It is hypothesized that the veterans who receive art therapy with CPT will show a significantly greater decrease in PTSD symptoms than those who receive only CPT.

ELIGIBILITY:
Inclusion Criteria:

* PCL-M initial score >= 50;
* Both genders,
* All ethnicities,
* Veterans in treatment for PTSD,

Exclusion Criteria:

* No active substance use disorder,
* No active suicidal or homicidal ideation,
* No psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-02-03 (Actual); Study Completion 2017-02-13 (Actual)

PRIMARY OUTCOMES:
PTSD Symptoms assessed by PCL-M score | 8-12 weeks
  PTSD symptoms will be measured by PCL-M score
Depression Symptoms assessed by Beck Depression Inventory-II | 8-12 weeks
  Beck Depression Inventory-II will be used to measure depression

SECONDARY OUTCOMES:
Treatment Satisfaction assessed by Likert scale | 8-12 weeks
  Likert scale will be used to compare satisfaction with art and CPT conditions
Treatment completion assessed by dropout rate | 8-12 weeks
  Compare dropout rate between experimental and control groups during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Cross, Ph.D., FNP, Study Chair — IRB Chair
Locations (1):
- Hampton VA Medical Center, Hampton, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be made available to other researchers. Aggregated data and de-identified data could be potentially be shared at a future date.